CLINICAL TRIAL: NCT01638377
Title: A Multi-site Study to Disseminate and Evaluate Pharmacotherapy for Alcohol Dependence in Convicted Drinking Drivers
Brief Title: Pharmacotherapy for Alcohol Dependence in Convicted Drinking Drivers
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment proved to be extremely difficult.
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Bernard Le Foll, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 079/2011
Record Dates: First submitted 2012-06-28; First posted 2012-07-11 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-04

CONDITIONS: Alcohol Dependence
Keywords: Back on Track; convicted drinking drivers; naltrexone; alcohol dependence
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naltrexone (Experimental): Drug: Naltrexone 50 mg/day for 24 weeks.All participants will receive medical intervention in the form of medical management (MM) which will be delovered by a trained health care professional.
  Interventions: Drug: Naltrexone
- Control (Placebo Comparator): Drug: Control Placebo (Lactose Monohydrate) for 24 weeks. All participants will receive medical intervention in the form of medical management (MM) which will be delivered by a trained health care professional.
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Naltrexone — 50 mg/day for 24 weeks. All participants will receive medical intervention in the form of medical management (MM) which will be delivered by a trained health care professional.
  Other Names: Revia
  Arms: Naltrexone
Drug: Control — Placebo (Lactose Monohydrate) for 24 weeks. All participants will receive medical intervention in the form of medical management (MM) which will be delivered by a trained health care professional.
  Other Names: Placebo (Lactose Monohydrate)
  Arms: Control

SUMMARY:
This pilot study will explore the ways to link Ontario's remedial system for convicted drinking drivers to medical intervention, assess the receptiveness of the Back on Track client population to effective medical interventions, and assess the feasibility of a full-scale trial of pharmacotherapy for convicted drinking drivers.

DETAILED DESCRIPTION:
Many individuals with Alcohol Dependence do not receive treatment, despite effective treatments being available. A significant healthcare challenge is to find ways to bring people who have alcohol dependence into treatment programs. Drinking drivers are a group that has been shown to have high rates of alcohol dependence. In Ontario, all convicted drinking drivers who want to obtain a drivers license must complete Ontario's remedial program for convicted drinking drivers called Back on Track (BOT). In this program, those with more serious alcohol-related problems are assigned to a group treatment program. While it is likely that many of the individual in this group are experiencing alcohol dependence, currently there is no formal linkage to any medical services for these problems. In this study, the investigators will provide those in the BOT treatment group with information about a 24-week study assessing the effectiveness of naltrexone vs. placebo. This study will also assess the feasibility and level of interest among this population to obtain treatment for alcohol dependence.

ELIGIBILITY:
Inclusion Criteria:

* Male or females - 18 years or older
* Been convicted of drinking driving and allocated to either the education or the treatment group of the BOT program
* Meet criteria for alcohol dependence using the SCID-IV
* Consume more than 14 drinks (female) or 21 drinks (male) per week with a minimum of 2 heavy drinking days (≥ 4 drinks for females and ≥ 5 drinks for males) during a consecutive 30-day period within the 90 days prior to the baseline evaluation
* Willing to receive pharmacotherapy for their alcohol dependence
* Seeking abstinence from alcohol as their main goal

Exclusion Criteria:

* History of other substance use (other than nicotine or cannabis) by DSM-IV criteria in the last 90 days (6 months for opiate abuse)
* Positive urine drug screen
* Psychiatric disorder requiring medication
* Unstable medical condition requiring immediate investigation or treatment
* Pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Participation rate | 2 years
  We will determine what percentage of subjects will participate in the preliminary medical screening and what percentage of subjects with a diagnosis of alcohol dependence will participate in the trial.

SECONDARY OUTCOMES:
Effect of naltrexone on drinking patterns and drinking related measures | At baseline and six-month follow-up
  Clinical trial data of naltrexone vs. placebo will assess the effectiveness of the study intervention on alcohol related outcomes. Outcomes will include percent days abstinent, time to first heavy drinking day and alcohol craving. BOT program data for all participants will also be assessed including measures of drinking behaviour and measures of other drug use and consequences resulting from substance use. Ministry of Transportation data will be used to determine the long term effect on relevant outcomes such as collisions and charges associated with alcohol use.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Le Foll, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Background] Anton RF, O'Malley SS, Ciraulo DA, Cisler RA, Couper D, Donovan DM, Gastfriend DR, Hosking JD, Johnson BA, LoCastro JS, Longabaugh R, Mason BJ, Mattson ME, Miller WR, Pettinati HM, Randall CL, Swift R, Weiss RD, Williams LD, Zweben A; COMBINE Study Research Group. Combined pharmacotherapies and behavioral interventions for alcohol dependence: the COMBINE study: a randomized controlled trial. JAMA. 2006 May 3;295(17):2003-17. doi: 10.1001/jama.295.17.2003. PMID 16670409
- [Background] Lee JD, Grossman E, DiRocco D, Truncali A, Hanley K, Stevens D, Rotrosen J, Gourevitch MN. Extended-release naltrexone for treatment of alcohol dependence in primary care. J Subst Abuse Treat. 2010 Jul;39(1):14-21. doi: 10.1016/j.jsat.2010.03.005. Epub 2010 Apr 2. PMID 20363090
- [Background] Lapham SC, Smith E, C'de Baca J, Chang I, Skipper BJ, Baum G, Hunt WC. Prevalence of psychiatric disorders among persons convicted of driving while impaired. Arch Gen Psychiatry. 2001 Oct;58(10):943-9. doi: 10.1001/archpsyc.58.10.943. PMID 11576032
- [Background] Mann RE, Anglin L, Wilkins K, Vingilis ER, MacDonald S. Mortality in a sample of convicted drinking drivers. Addiction. 1993 May;88(5):643-7. doi: 10.1111/j.1360-0443.1993.tb02076.x. PMID 8518714
- [Background] Impinen A, Makela P, Karjalainen K, Rahkonen O, Lintonen T, Lillsunde P, Ostamo A. High mortality among people suspected of drunk-driving. An 18-year register-based follow-up. Drug Alcohol Depend. 2010 Jul 1;110(1-2):80-4. doi: 10.1016/j.drugalcdep.2010.02.007. Epub 2010 Mar 23. PMID 20334987
- [Background] COMBINE Study Research Group. Testing combined pharmacotherapies and behavioral interventions in alcohol dependence: rationale and methods. Alcohol Clin Exp Res. 2003 Jul;27(7):1107-22. doi: 10.1097/00000374-200307000-00011. PMID 12878917
- [Background] Rosner S, Hackl-Herrwerth A, Leucht S, Vecchi S, Srisurapanont M, Soyka M. Opioid antagonists for alcohol dependence. Cochrane Database Syst Rev. 2010 Dec 8;(12):CD001867. doi: 10.1002/14651858.CD001867.pub3. PMID 21154349
- [Background] Sullivan JT, Sykora K, Schneiderman J, Naranjo CA, Sellers EM. Assessment of alcohol withdrawal: the revised clinical institute withdrawal assessment for alcohol scale (CIWA-Ar). Br J Addict. 1989 Nov;84(11):1353-7. doi: 10.1111/j.1360-0443.1989.tb00737.x. PMID 2597811
- [Background] Sobell LC, Sobell MB, Leo GI, Cancilla A. Reliability of a timeline method: assessing normal drinkers' reports of recent drinking and a comparative evaluation across several populations. Br J Addict. 1988 Apr;83(4):393-402. doi: 10.1111/j.1360-0443.1988.tb00485.x. No abstract available. PMID 3395719
- [Background] Tonigan JS, Miller WR, Brown JM. The reliability of Form 90: an instrument for assessing alcohol treatment outcome. J Stud Alcohol. 1997 Jul;58(4):358-64. doi: 10.15288/jsa.1997.58.358. PMID 9203116
- [Background] Rollnick S, Heather N, Gold R, Hall W. Development of a short 'readiness to change' questionnaire for use in brief, opportunistic interventions among excessive drinkers. Br J Addict. 1992 May;87(5):743-54. doi: 10.1111/j.1360-0443.1992.tb02720.x. PMID 1591525
- [Background] MacKillop J. Factor structure of the alcohol urge questionnaire under neutral conditions and during a cue-elicited urge state. Alcohol Clin Exp Res. 2006 Aug;30(8):1315-21. doi: 10.1111/j.1530-0277.2006.00159.x. PMID 16899034
- [Background] Drummond DC, Phillips TS. Alcohol urges in alcohol-dependent drinkers: further validation of the Alcohol Urge Questionnaire in an untreated community clinical population. Addiction. 2002 Nov;97(11):1465-72. doi: 10.1046/j.1360-0443.2002.00252.x. PMID 12410786
- [Background] HAMILTON M. The assessment of anxiety states by rating. Br J Med Psychol. 1959;32(1):50-5. doi: 10.1111/j.2044-8341.1959.tb00467.x. No abstract available. PMID 13638508
- [Result] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- See also: Information about research at the Centre for Addiction and Mental Health — http://www.camh.net/research